CLINICAL TRIAL: NCT05775835
Title: Effects of Whole Body Vibration and Resistance Exercise on Carotis Intima Media Thickness and Muscle Architecture in Patients With Hypertension
Brief Title: Effects of Whole Body Vibration and Resistance Exercise on Carotis Intima Media and Muscle Architecture in Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Collaborators: Health Institutes of Turkey (Other Government)
Responsible Party: Principal Investigator, Menekse Safak, Res. Assist., Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS2022/032
Record Dates: First submitted 2023-02-13; First posted 2023-03-20 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2023-07

CONDITIONS: Hypertension; Whole Body Vibration; Muscle Architecture; Carotid Intima Media Thickness
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Whole body vibration exercise group (Experimental): The application will be carried out with a whole body vibration device that gives 35 Hz constant vertical vibration. The exercises will be performed on the vibration platform in a standing position and with vibration. 5 static squats (in 90 degrees knee extension), mini squats (120 degrees knee extension), mini squat on the fingertip (120 degrees knee extension), right and left lunge positions, which will be accepted as 180 degrees full knee extension exercise protocol. During the squat exercises, the patient will be positioned with their feet open at shoulder level and the knee flexion angle will be adjusted with a goniometer by the physiotherapist before each training session. For static exercises, the duration will be 3 sets of 30-60 seconds in each practice position. There will be 30-60 second rest breaks between sets.
  Interventions: Other: Whole body vibration exercise
- Strength training group (Experimental): The exercises will be performed on the vibration platform but without vibration. Patients will be asked to hold a "body bar" corresponding to 10% of their body weight during exercises. 5 dynamics including squats (in 90 degrees knee extension), mini squats (120 degrees knee extension), mini squats on the toe tip (120 degrees knee extension), right and left lunge exercises, which will be accepted as 180 degrees full knee extension will perform an exercise protocol consisting of exercise. During the squat exercises, the patient will be positioned with their feet open at shoulder level and the knee flexion angle will be adjusted with a goniometer by the physiotherapist before each training session. For dynamic exercise, the duration will be 3 sets of 10 repetitions. Dynamic exercises will be performed with slow and controlled movements, consisting of 3 seconds of eccentric and 2 seconds of concentric phases.
  Interventions: Other: Strengthening exercise
- Whole body vibration and strengthening exercise group (Experimental): In the TVVE+KE group, the selected exercises will be performed with vibratory and dynamic strengthening exercises on the vibration platform. The application will be carried out on a whole body vibration device giving a constant vibration of 35 Hz. Patients will be asked to hold a "body bar" corresponding to 10% of their body weight during exercises. 5 dynamics including squats (in 90 degrees knee extension), mini squats (120 degrees knee extension), mini squats on the toe tip (120 degrees knee extension), right and left lunge exercises, which will be accepted as 180 degrees full knee extension will perform an exercise protocol consisting of exercise. D For dynamic exercise, the duration will be 3 sets of 10 repetitions. Dynamic exercises will be performed with slow and controlled movements, consisting of 3 seconds of eccentric and 2 seconds of concentric phases.
  Interventions: Other: Whole body vibration and strengthening exercise
- Control Group (No Intervention): No exercise recommendations or interventions will be made to the patients in the control group.

INTERVENTIONS:
Other: Whole body vibration and strengthening exercise — Prior to commencing training, all subjects will undergo a pre-screening that includes a thorough history and physical examination to monitor compliance with the inclusion criteria. Evaluation parameters will be evaluated before and after 6 weeks of exercise. Training sessions will be held 3 days a week for 6 weeks, with a minimum of 48 hours between training sessions. All exercise groups include a warm-up period and a cool-down period (stretching exercises). Stretching exercises for the hamstring, gastrocnemius, soleus, and quadriceps muscles will be performed for 15-30 seconds and 3-5 repetitions. The total average application time (including warm-up and cool-down exercises), consisting of exercise and rest periods, was planned as 45-60 minutes for the WBV, SE, and WBV+SE groups.
  Arms: Whole body vibration and strengthening exercise group
Other: Whole body vibration exercise — The application will be carried out with a whole body vibration device that gives 35 Hz constant vertical vibration. The exercises will be performed on the vibration platform in a standing position and with vibration. 5 static squats (in 90 degrees knee extension), mini squats (120 degrees knee extension), mini squat on the fingertip (120 degrees knee extension), right and left lunge positions, which will be accepted as 180 degrees full knee extension exercise protocol. During the squat exercises, the patient will be positioned with their feet open at shoulder level and the knee flexion angle will be adjusted with a goniometer by the physiotherapist before each training session. For static exercises, the duration will be 3 sets of 30-60 seconds in each practice position. There will be 30-60 second rest breaks between sets.
  Arms: Whole body vibration exercise group
Other: Strengthening exercise — The exercises will be performed on the vibration platform but without vibration. Patients will be asked to hold a "body bar" corresponding to 10% of their body weight during exercises. 5 dynamics including squats (in 90 degrees knee extension), mini squats (120 degrees knee extension), mini squats on the toe tip (120 degrees knee extension), right and left lunge exercises, which will be accepted as 180 degrees full knee extension will perform an exercise protocol consisting of exercise. During the squat exercises, the patient will be positioned with their feet open at shoulder level and the knee flexion angle will be adjusted with a goniometer by the physiotherapist before each training session. For dynamic exercise, the duration will be 3 sets of 10 repetitions. Dynamic exercises will be performed with slow and controlled movements, consisting of 3 seconds of eccentric and 2 seconds of concentric phases.
  Arms: Strength training group

SUMMARY:
Exercise is of great importance in the treatment of hypertension, which is expressed as a very serious disease, the prevalence of which is increasing day by day in the world and can cause many complications that are common in society. Exercise methods effective on carotid intima-media thickness, skeletal muscle architecture, and strength, which are important markers of hypertension-related organ damage, remain unclear. Strengthening exercises draw attention as an important approach in the control of hypertension. In order for strengthening exercises to be effective in the rehabilitation of hypertension, moderate and high-intensity exercises are recommended. New exercise approach strategies are gaining importance in order to enable resistance exercise training and to increase muscle mass and strength in the elderly who have a limitation for the recommended exercise intensity, in patients with hypertension, and in people with various diseases in which the cardiovascular system is affected. Whole body vibration (TVV) applications, which have no side effects reported as the current example of these exercise approaches, attract attention. Many positive effects occur on the cardiovascular system with the short-term and low-effort application of TVV exercise approaches, which are frequently used in routine rehabilitation practices. However, when the literature is examined, the effects of these exercise approaches on carotid intima-media thickness, which is one of the main markers of hypertension-related organ damage, are unclear. In addition, the effects of hypertension on quadriceps muscle architecture, which are expected to be adversely affected as a result of affecting autophagy regulation in skeletal muscle and causing decreased muscle capillarization, remain unclear. In addition, there is insufficient data on the effectiveness of strengthening exercises and TVV exercises on hemodynamic responses and quadriceps muscle strength in hypertensive patients. It will shed light on the determination of the exercise approach that is most effective on the muscle architecture, hemodynamic responses and carotid intima-media thickness of hypertensive patients and that can show these effects without overloading the cardiovascular system.

DETAILED DESCRIPTION:
Hypertension is a very serious disease that can cause many complications such as stroke, coronary heart disease, heart failure, kidney failure, and visual impairment, which is more common in the world. Hypertension-related organ damage (i.e. increased left ventricular mass index, left atrial dilatation, left ventricular dysfunction, carotid thickening and/or plaque, increased arterial stiffness, decreased glomerular filtration rate, and urinary albumin excretion), which is one of the key parameters in linking hypertension with many diseases, It is considered a strong predictor of cardiovascular disease. As a result of organ damage associated with hypertension, various changes are encountered in the skeletal and cardiac muscle and vascular structure. The importance of autophagy regulation specific to skeletal muscle is known in the structure of skeletal muscle. It has been reported that hypertension affects autophagy regulation in skeletal muscle, causing a decrease in type I fiber percentage and size, altered contractive function, and high apoptotic signaling. Numerous studies have demonstrated an association between vascular status and skeletal muscle health.In hypertensive patients, the presence of some degenerated capillaries adjacent to the muscle fibers is interpreted as the beginning of a process of degeneration and reduction in capillarization. With hypertension, capillaries show morphological changes and the wall thickness/lumen ratio increases. It is stated that with hypertension, muscle capillarization and oxygenation decrease and arterial dysfunction in the lower extremities causes decreases in muscle strength. Considering the data in the literature, it is thought that patients with hypertension may encounter changes in muscle architecture. Skeletal muscle architecture (including muscle cross-sectional area, thickness, and angle of fascicle pennation) are key determinants of a muscle's maximum strength.A tendency to decrease in quadriceps strength has been described in patients with hypertension. It is thought that this adaptation is probably related to local changes in the fiber type ratio and area of the VL muscle rather than a systemic adaptation. In addition, a tissue-specific effect of angiotensin II in skeletal muscle cell has been described. Accordingly, the release of angiotensin II appears to contribute to an increase in the lactate/pyruvate ratio caused by an impairment in glucose supply to skeletal muscle. As a result, hypertension can cause muscle disuse and deterioration of functional capacity. An increase in carotid intima-media thickness (CIMT), one of the markers of hypertension-related organ damage, also occurs as a result of changes in cardiac and vascular structures seen as a result of hypertension. Reversal or reduction of target organ damage is a valuable parameter in the evaluation of antihypertensive therapy efficacy, as regression of cardiac and vascular changes has been shown to be associated with improved prognosis for long-term cardiovascular events. It is important to determine the necessary treatment approaches to control and reduce these negative changes observed in hypertensive patients.

Today, lifestyle modifications such as increasing physical activity and regulating nutrition, as well as antihypertensive drugs, come to the fore in the treatment of hypertension. Regular exercise has a protective effect in the prevention, treatment and control of hypertension. Regular exercise as a part of lifestyle change seems to be as effective as drugs in the treatment of hypertension. With regular exercise, an average of 5 mmHg reduction in blood pressure can be achieved. With a 5 mmHg decrease in systolic blood pressure, death due to coronary heart disease decreases by 9%, death due to stroke by 14%, and death due to all causes by 7%. Muscle capillary enlargement and thus an increased capillary density have also been reported in hypertensive patients with exercise training. Considering these reasons, regular exercise should be recommended for all individuals, including normotensives, prehypertensives and hypertensives.

The importance of strength training, like many exercise approaches, in reducing resting blood pressure in hypertensive patients is known. It has been reported that a significant reduction in systolic and diastolic blood pressures was observed in all of the quadriceps, latissimus dorsi and biceps muscles after strengthening exercises and compared to resting pressure levels at different exercise intensities. Additionally, it has been shown that the change in blood pressure is greater when strengthening exercise is given to the quadriceps muscle. Resistant arterial hypertension can cause muscle disuse and decrease in functional capacity due to arterial and target organ lesions. In addition to the cardiovascular effects of strengthening exercises, the effects of increasing muscle strength and reducing high blood pressure observed during exercise have been reported. It has been stated that the strengthening exercise program given for the quadriceps in patients with resistant hypertension effectively increases the quadriceps muscle strength by increasing the maximum isometric contraction values of the vastus lateralis and vastus medialis without adversely affecting the cardiovascular variables. In another study, a decrease in the waist circumference, pre-peritoneal (visceral) and thigh fat thickness, and an increase in the thigh muscle thickness were reported in exercises such as squats and taking a step forward for 12 weeks.Strengthening exercises are known to be effective in increasing rectus femoris muscle thickness and muscle strength in overweight or obese women with metabolic syndrome, but there is a lack of literature on the effect of strengthening exercises on muscle architecture in hypertensive patients. The increase in carotid intima-media thickness, which is one of the important markers associated with hypertension, is due to thickening of the intima and/or media layer. Atherosclerosis, which is primarily caused by endothelial dysfunction, is responsible for intimal thickening, and smooth muscle hypertrophy, usually due to hypertension, is responsible for median thickening. Strengthening exercises combined with aerobic exercise are known to be effective in reducing carotid intima-media thickness in overweight and obese, young and old women. In addition, a relationship has been shown between the change in carotid intima-media thickness and walking speed, which is one of the parameters of the functional level. It is known that regular exercise also delays carotid intima-media thickness in hypertensive patients, but the effects of strengthening exercise on carotid intima-media thickness in hypertensive patients are unclear.

It is recommended that the strengthening exercise, which should be planned to increase muscle strength in hypertensive patients, should be at an intensity of 70% of 1 maximum repetition on average. However, people with cardiovascular diseases or hypertension may be at risk of overloading the cardiovascular system and an increased risk of cardiac events when performing high-intensity resistance exercises. New exercise approach strategies are gaining importance in order to enable resistance exercise training and to increase muscle mass and strength in the elderly who have a limitation for the recommended exercise intensity, in patients with hypertension, and in people with various diseases in which the cardiovascular system is affected. A current example of these exercise approaches are exercises with whole body vibration. Whole body vibration (WBV) exercises are a new exercise training option that can reduce the time and effort required to achieve significant musculoskeletal and cardiovascular system gains. WBV exercises are performed while standing on a platform that creates repeated and rapid swings and supports automatic body adaptations. These dynamic oscillations provide repeated and intense eccentric-concentric muscle contractions that reinforce the normal muscle contractions performed. Adding whole body vibration application to strengthening exercises increases the oxygen demand of the muscle during exercise. In a study evaluating the acute effects of whole-body vibration in prehypertensive patients, it was reported that whole-body vibration applications combined with resistance exercise increased post-exercise hypotension responses and post-exercise oxygen consumption more.Alternatively, whole body vibration exercise (WBV) training is known to be a potential rehabilitation method for muscle and artery function. It has been reported that whole body vibration exercise training in postmenopausal hypertensive women reduces cardiovascular risks by improving aortic wave reflection, muscle strength, systemic and leg arterial stiffness. In another study, it was stated that 8-week whole body vibration training was effective in improving semoatovagal balance and blood pressure. It is predicted that when the body is exposed to vibration, it induces rhythmic muscle contractions that can cause changes in peripheral arteries. The expansion of capillaries in the muscles facilitates the exchange of nutrients, metabolic byproducts and oxygen between cells and capillaries. Whole body vibration applications are promising in the treatment of deterioration in muscle architecture, which can be seen as a result of decreased muscle capillarization and oxygenation associated with hypertension. In a study examining the effects of 6-week whole body vibration and traditional strengthening exercises on vascular adaptation in healthy adults, it was shown that whole body vibration was effective in reducing carotid intima-media thickness. However, the effect of whole body vibration on carotid intima-media thickness, which is also an indicator of arterial stiffness, is unclear in hypertensive patients. It has been shown that WBV exercises have similar effects on muscle strength and arterial stiffness as strengthening exercises in a wide range of populations, with the greatest effect in elderly individuals with limited muscle function. Similarly, there are various studies showing the effect of whole body vibration exercises on muscle strength and muscle architecture in different patient groups, but the literature on the effectiveness in hypertensive patients is insufficient.

When the data in the literature is examined, the importance of determining the effects of whole body vibration and strengthening exercises on carotid intima media thickness and muscle architecture in hypertensive patients draws attention. In our study, it is aimed to determine the effects of whole body vibration (WBV) and strengthening exercises (SE) on hemodynamic responses, carotid intima-media thickness, quadriceps muscle strength and architecture in hypertensive patients in the light of information in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 30-59,
* Being diagnosed with stable hypertension in stage 1 (systolic blood pressure 140-159 mmHg and diastolic blood pressure 90-99 mmHg) and stage 2 (systolic blood pressure 160-179 mmHg and diastolic blood pressure 100-109 mmHg),
* Not being obese (BMI<30 kg/m2)
* Not having the habit of exercise (regular exercise <60 min/week or not doing any strengthening exercise),
* Not having a history of smoking,
* Volunteering to participate in the study

Exclusion Criteria:

* Having any additional disease other than hypertension, such as diabetes mellitus, heart failure, unstable angina, myocardial infarction, kidney disease and psychiatric disease related to circulatory, orthopedic, neurological, cardiac and respiratory functions,
* Using hormonal supplements,
* Hypertension-related medication change in the last 4 weeks

Ages: 30 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Carotid intima media thickness | Change from Baseline Carotid Intima Media Thickness at 6 weeks
  Carotid intima-media thickness (CIMT) is an independent marker of the onset of hypertension. It is also known that there is a close relationship between carotid intima media thickness and blood pressure.Carotid artery B-Mode ultrasonography examinations in the evaluation of carotid intima-media thickness EPIQ Elite Diagnostic Ultrasound System Release 7.0.5. It will be done with L18-4 MHz linear transducer using Philips ultrasonography device.
Quadriceps muscle architecture-muscle thickness | Change from Baseline Muscle Thickness at 6 weeks
  Muscle architecture including rectus femoris, vastus lateralis, vastus medialis oblique and vastus intermedius muscle thicknesses will be evaluated.Maximal muscle thickness will be measured as the distance between the superficial and deep fascia at the widest distance on transversal views.All images will be taken by the same investigator and from the same anatomical region.Muscle architecture examination will be performed using the Philips ultrasonography system.
Quadriceps muscle architecture-pennation angle | Change from Baseline Pennation Angle at 6 weeks
  Muscle architecture including vastus lateralis and vastus medialis oblique pennation angles will be evaluated.Pennation angle is defined as the angle between the muscle fibers and the deep fascia of the muscle. Therefore, pennation angles will be measured on the longitudinal ultrasound image. Since the orientation of the rectus femoris and vastus intermedius fibers is almost parallel to their fascia, the angle of pennation for these muscles of the quadriceps muscle was not determined. All images will be taken by the same investigator and from the same anatomical region. Muscle architecture examination will be performed using the Philips ultrasonography system.
Quadriceps muscle architecture-muscle cross-section area | Change from Baseline Muscle Cross-section Areas at 6 weeks
  Muscle architecture including rectus femoris, vastus lateralis, vastus medialis oblique and vastus intermedius muscle cross-section areas will be evaluated.Muscle cross-sectional area measurement will be calculated by drawing the boundaries of the muscle through a program in the ultrasound device. All images will be taken by the same investigator and from the same anatomical region. Muscle architecture examination will be performed using the Philips ultrasonography system.
Lower extremity muscle strength | Change from Baseline Lower Extremity Muscle Strength at 6 weeks
  The isometric muscle strength of the quadriceps muscles of the individuals participating in our study will be evaluated using a portable hand dynamometer (Lafayette Manual Muscle Tester, model 01163, USA).
Hemodynamic responses- blood pressure change | Change from Baseline Systolic Blood Pressure and Diastolic Blood Pressure at 6 weeks.
  Systolic blood pressure values and diastolic blood pressure values will be noted separately. A digital blood pressure monitor will be used to assess blood pressure.
Hemodynamic responses-saturation | Change from Baseline Saturation at 6 weeks
  Saturation (oxygen carrying capacity (SpO2)) will be evaluated with a finger-mounted portable pulse oximeter device.
Hemodynamic responses-heart rate | Change from Baseline Heart Rate at 6 weeks
  A digital heart rate monitor (Polar watch) will be used for heart rate.
Hemodynamic responses-respiratory frequency | Change from Baseline Respiratory Frequency at 6 weeks
  Respiratory frequency will be calculated by counting the breaths taken by the patient for 1 minute with a stopwatch.

SECONDARY OUTCOMES:
Hemodynamic responses- blood pressure | pre-intervention and immediately after the intervention
  Hemodynamic responses will be evaluated before and after exercise to monitor possible complications. blood pressure values and diastolic blood pressure values will be noted separately. A digital blood pressure monitor will be used to assess blood pressure.Assessment will be performed after the patient has rested in a sitting position for at least 5 minutes, immediately after exercise, and 3 minutes after exercise (after recovery).
Hemodynamic responses- heart rate | pre-intervention and immediately after the intervention
  Hemodynamic responses will be evaluated before and after exercise to monitor possible complications.Assessment will be performed after the patient has rested in a sitting position for at least 5 minutes, immediately after exercise, and 3 minutes after exercise (after recovery).
Hemodynamic responses-saturation | pre-intervention and immediately after the intervention
  Hemodynamic responses will be evaluated before and after exercise to monitor possible complications.Assessment will be performed after the patient has rested in a sitting position for at least 5 minutes, immediately after exercise, and 3 minutes after exercise (after recovery).
Hemodynamic responses-respiratory frequency | pre-intervention and immediately after the intervention
  Hemodynamic responses will be evaluated before and after exercise to monitor possible complications.Assessment will be performed after the patient has rested in a sitting position for at least 5 minutes, immediately after exercise, and 3 minutes after exercise (after recovery).

CONTACTS AND LOCATIONS:
Locations (1):
- Süleyman Demirel Universty, Isparta, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No